CLINICAL TRIAL: NCT06043570
Title: Evaluation of Clinical and Economic Benefit Using Remote Monitoring in Patients With Pacemaker (REMOTE-PM)
Brief Title: Benfit of Remote Monitoring in Pacemaker
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1-2022-0049
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Pacemaker Implanted Patients
Keywords: Pacemaker; remote monitoring; benefit, economic; financial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Monitoring follow up (Experimental)
  Interventions: Device: Remote Monitoring arm
- Conventional Follow up (No Intervention)

INTERVENTIONS:
Device: Remote Monitoring arm — Patients will be follow-up using remote monitoring. In the RM follow-up arm, the patients are not mandated to visit the clinic unless there is unscheduled call due to adverse event notification.
  Arms: Remote Monitoring follow up

SUMMARY:
Modern CIEDs are equipped with remote monitoring (RM) technology, which provides automatic transmissions of diagnostics and technical data from the implanted devices to the attending physician. RM has been shown to be a safe alternative to the conventional in-hospital visits, especially for low-risk patients, such as pacemaker recipients. These regular office visits include examinations of device function and patient clinical status, and may prompt the reprogramming of the device or changes in medication regimens. The efficiency of this strategy is, however, questionable since, in the majority of scheduled visits, the device programming or drug regimen is left unchanged. To optimize the follow-up of device recipients, systems have been developed, which allow the automatic teletransmission of data stored in the devices' memories, including battery voltage, lead characteristics, and arrhythmias. The data sent by a home transmitter allow the remote surveillance of patients and eliminate unnecessary ambulatory visits. Clinical studies of these new systems have been conducted mostly in recipients of cardioverter defibrillators, and only a few studies of permanently paced patients have been published.

However, due to the absence of medical regulations and systems for remote monitoring in Korea, the government does not provide clear guidelines and the Korean HIRA (Health Insurance Review & Assessment Service) is yet to set any reimbursement standards for home-transmitter and remote monitoring. As a result, most Korean physicians cannot practically use remote monitoring for CIED patients. Therefore, this project shall contribute to address the benefits of remote monitoring to the government and expediate the system to be set in the country.

Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia in the general population. AF has enormous socioeconomic implications because it increases the risk of mortality and morbidity resulting from stroke, congestive heart failure, dementia and impaired quality of life. To prevent the AF-related complication, early detection of AF is very important. Despite the latest HRS Expert Consensus Statement which has set a class I recommendation for RM as useful tool for the early detection and quantification of AF, there are still few data on the clinical reactions triggered by the AHRE detected by RM of CIEDs and on their possible benefit on patient's outcome.

The incidence of atrial high rate episodes (AHRE)/subclinical AF in patients with a pacemaker/implanted device is 30-70%, but it may be lower in the general population. Longer episodes of AHRE/subclinical AF (minimum of 5-6 min) are associated with an increased risk of clinical AF, ischemic stroke, major adverse cardiovascular events, and cardiovascular death.13 Clinical AF will reportedly develop in 1 in 5-6 of patients within 2.5 years after diagnosing AHRE/subclinical AF.

The remote monitoring feature is available in all geographies while it is yet to be reimbursed in South Korea. To be reimbursed by the NHIS of Korea, the data supporting the benefit of RM is necessary. By comparing clinical and economic benefits of remote monitoring, we might be able to set a guideline on the usage of remote monitoring in pacemaker patients.

DETAILED DESCRIPTION:
* Study Objective Primary study objective The primary objective of this non-inferiority, prospective trial in Korean population is to confirm that the proportion of patients who experienced at least one major adverse event (MAE), including (i) death, (ii) hospitalization for complications related to the pacing system, and (iii) hospitalization for an adverse cardiovascular event, is not higher in the remote follow-up (active) than in the standard care (control) group.
* Secondary objectives The secondary objectives of the trial are to address the economic benefits of remote monitoring to the government and expediate the system to be set in the country. Through this trial, we expect to set reimbursement policy in corporation with KHRS (Korean Heart Rhythm Society) including home transmitter. In addition, since Korea has one of the highest usage rate of smartphones even in elderly groups compared to Europe or North America, we are to suggest a set of guidelines for patient care and follow up schedules for remote monitoring patients according to Korean culture and circumstances.
* Study Design We propose to prospectively recruit 900 patients with pacemaker with SenseAbility feature implantation in multiple sites in Korea.

  * Eligible patients should be enrolled in remote monitoring system 0 to 45 days after successful device implantation and then randomly assigned in a 1:1 ratio to the RM or conventional follow-up group.
  * In the RM follow-up arm, the patients are not mandated to visit the clinic unless there is unscheduled call due to adverse event notification.
  * In the conventional follow-up arm, the patients should be seen at the clinic according to each center's custom but no longer than 1 year between each visit. Follow-up should be continued accordingly until two-years of device implant.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years

  * Patients with permanent pacemaker with SenseAbility feature & RM

    * Ability to provide informed consent and to complete the study and required follow-up ④ Those who refuse to use remote monitoring system or who live in an environment where remote monitoring system cannot be utilized.

      * Patient who refuse to use or expected to use less than 75% of remote monitoring system.

Exclusion Criteria:

* Severe hepatic and renal insufficiency (AST or ALT ≥ three times of normal upper limit; SCr > 3.5 mg/dl or Ccr < 30ml/min)

  * Thyroid gland dysfunction

    * Pregnancy ④ Malignant tumor

      * Severe organic heart disease (such as moderate to severe mitral regurgitation, dilated cardiomyopathy, hypertrophic cardiomyopathy, severe heart valve disease)

        * Life expectancy < 12 months ⑦ Patients unable or unwilling to cooperate in the study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
major adverse event (MAE) | Arm 1: 6 month, 12 month, 18 month, 24 month, anytime using remote monitoring - Arm 2: 6 month, 12 month, 18 month, 24 month
  major adverse event (MAE), including all-cause death and hospitalizations for device-related or cardiovascular adverse events

SECONDARY OUTCOMES:
Economic benefit by remote mononitoring | 24 month
  economic benefit of each treatment
all-cause death | Arm 1: 6 month, 12 month, 18 month, 24 month, anytime using remote monitoring - Arm 2: 6 month, 12 month, 18 month, 24 month
hospitalizations for device-related events | Arm 1: 6 month, 12 month, 18 month, 24 month, anytime using remote monitoring - Arm 2: 6 month, 12 month, 18 month, 24 month
cardiovascular adverse events | Arm 1: 6 month, 12 month, 18 month, 24 month, anytime using remote monitoring - Arm 2: 6 month, 12 month, 18 month, 24 month
AHRE/subclinical AF | Arm 1: 6 month, 12 month, 18 month, 24 month, anytime using remote monitoring - Arm 2: 6 month, 12 month, 18 month, 24 month
clinical AF | Arm 1: 6 month, 12 month, 18 month, 24 month, anytime using remote monitoring - Arm 2: 6 month, 12 month, 18 month, 24 month
time to change of management including OAC | Arm 1: 6 month, 12 month, 18 month, 24 month, anytime using remote monitoring - Arm 2: 6 month, 12 month, 18 month, 24 month

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No